CLINICAL TRIAL: NCT00742898
Title: Non-targeted Opt-out Rapid HIV Screening in the Emergency Department: a Controlled Clinical Trial
Brief Title: Evaluation of Opt-Out Rapid HIV Testing in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Jason S. Haukoos, MD, MSc / Director of Emergency Medicine Research, Denver Health Medical Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 06-0820; U18PS000314 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-08-28 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: HIV Infections
Keywords: Quasi-experimental design; Non-targeted opt-out rapid HIV screening; Diagnostic rapid HIV testing; Emergency department; Effectiveness; Efficiency; Health services research; Program evaluation; Effectiveness and efficiency of non-targeted rapid HIV screening in the ED
MeSH Terms: conditions — HIV Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Non-targeted opt-out rapid HIV screening fully integrated into an urban, inner-city ED.
  Interventions: Other: Non-targeted opt-out rapid HIV screening
- 2 (Active Comparator): Diagnostic rapid HIV testing fully integrated into an urban, inner-city ED.
  Interventions: Other: Non-targeted opt-out rapid HIV screening

INTERVENTIONS:
Other: Non-targeted opt-out rapid HIV screening — Experimental Arm: Integrated non-targeted opt-out rapid HIV screening Active Comparator Arm: Integrated diagnostic rapid HIV testing

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of performing opt-out rapid HIV screening in an urban, inner-city emergency department, as well as to evaluate its clinical efficiency, cost effectiveness, and patient and staff satisfaction.

DETAILED DESCRIPTION:
An estimated 40,000 new HIV infections occur annually in the United States. Although significant effort has been devoted to improving identification of patients with undiagnosed HIV infection, this rate has changed very little in the last decade and new infections appear to be increasing most in non-traditional risk groups, including racial and ethnic minorities. Most persons infected with HIV still do not get tested until late in their disease courses, primarily due to its long asymptomatic period and their relatively poor access to routine medical care. Over 100 million people visit emergency departments (EDs) annually, and the ED commonly serves as a patient's only source for medical care, and thus the only potential opportunity to receive HIV counseling, testing, and referral (CTR). Also, patients who are most likely to use the ED as their only source of care are often those for whom the HIV epidemic is spreading most. The primary objective of the proposed research is to demonstrate clinical effectiveness, clinical efficiency, cost effectiveness, and patient-staff satisfaction with performing routine voluntary opt-out rapid HIV CTR in a high-volume urban ED, when compared to a targeted rapid HIV CTR program in the same setting. The primary hypothesis of the proposed investigations is that opt-out rapid HIV CTR is associated with a higher rate of overall testing, identification of patients infected with HIV, identification of patients infected with HIV earlier in their disease courses, and successful linkage into medical and preventative care for those patients who test positive for HIV infection. The secondary hypotheses are that opt-out rapid HIV CTR: (1) is not associated with increased ED processes of care, defined by patient waiting times, length of stays, the proportion of patients who leave before completing their evaluations, and an overcrowding index; and (2) is cost-effective. The tertiary hypotheses are that opt-out rapid HIV CTR is associated with a higher level of patient and ED staff satisfaction. To address these hypotheses, we will perform a prospective quasi-experimental equivalent time-samples clinical trial in which consecutive patients who present to the ED during interventional periods will be offered opt-out rapid HIV CTR as part of their visits, and during the control periods, patients will be targeted by physicians for rapid HIV CTR using a previously developed and validated CTR model. The results obtained from this study will improve our understanding of how best to identify patients with HIV infection in ED, and whether opt-out rapid HIV CTR is an effective means to achieve the CDC's goals of identifying more asymptomatic HIV-infected patients earlier in their disease courses.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Emergency department patients

Exclusion Criteria:

* <16 years
* Unable to provide consent (e.g., intoxicated, altered mental status)
* Critical illness
* Prisoners or detainees
* Already known to be infected with HIV
* Victims of sexual assault
* Occupational exposures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120000 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
HIV seropositivity | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Jason S. Haukoos, MD, MSc, Principal Investigator — Denver Health Medical Center; Emily Hopkins, MSPH, Study Director — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Haukoos JS, Hopkins E, Byyny RL, Conroy AA, Silverman M, Eisert S, Thrun M, Wilson M, Boyett B, Heffelfinger JD; Denver ED HIV Opt-Out Study Group. Design and implementation of a controlled clinical trial to evaluate the effectiveness and efficiency of routine opt-out rapid human immunodeficiency virus screening in the emergency department. Acad Emerg Med. 2009 Aug;16(8):800-8. doi: 10.1111/j.1553-2712.2009.00477.x. PMID 19673717